CLINICAL TRIAL: NCT06403098
Title: The Effects of External Nasal Dilator Strips on Sleep and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Joseph Watso, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00004863
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No External Nasal Dilator Strip (No Intervention): The control arm will last 7 consecutive nights and days. Participants will be asked to follow normal activity and sleep patterns. Immediately after waking the participants will measure their blood pressure and heart rate variability and complete a sleep diary to characterize subjective sleep quality. A wrist-based activity monitor will measure objective sleep quality during the control arm.
- External Nasal Dilator Strip (Experimental): The experimental arm will last 7 consecutive nights and days. Participants will be asked to follow normal activity and sleep patterns, but they will wear an external nasal dilator strip during sleep. Immediately after waking the participants will measure their blood pressure and heart rate variability and complete a sleep diary to characterize subjective sleep quality. A wrist-based activity monitor will measure objective sleep quality during the experimental arm.
  Interventions: Device: External Nasal Dilator Strip

INTERVENTIONS:
Device: External Nasal Dilator Strip — Participants will wear an extra strength Breathe Right nasal strip overnight.
  Arms: External Nasal Dilator Strip

SUMMARY:
The goal of this interventional study is to learn if wearing an external nasal dilator strip while sleeping changes objective and perceived sleep quality, immediate post-waking blood pressure, and immediate-post waking heart rate variability.

DETAILED DESCRIPTION:
Nasal dilator strips are strips often made up of stiff plastic, placed on the lower bridge of the nose by an adhesive strip. They work by slightly pulling the nostrils and surrounding nose bridge area outward, dilating the nostrils, and decreasing air resistance. Nasal breathing is associated with lower diastolic blood pressure, an important marker of heart health, in comparison to mouth breathing. In addition to blood pressure, nasal breathing during sleep is potentially related with better sleep quality. Participating in this study will help us understand the effect nasal dilator strips have on cardiovascular and sleep health. Better understanding of the benefits of nasal dilator strips will provide important knowledge to researchers who study how the body works.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* BMI <30
* Has a smartphone and is willing to download EliteHRV and OMRON mobile applications.
* Able to use a nasal dilator strip

Exclusion Criteria:

* Overt cardiovascular (e.g., diagnosed hypertension), respiratory, neurological, renal, liver, and/or metabolic health conditions.
* Current or recent (regular use within the past 6 months) use of tobacco or nicotine products (e.g., cigarettes).
* Currently pregnant, trying to become pregnant, or lactating.
* Inability to breathe through the nose.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Weekly averaged systolic blood pressure | Immediate post-waking for 14 consecutive days. Weekly averages (e.g. day 1-7 vs 8-14) will be compared between conditions.
  Brachial systolic blood pressure will be measured with an automated blood pressure monitor (OMRON BP5250).
Weekly averaged diastolic blood pressure | Immediate post-waking for 14 consecutive days. Weekly averages (e.g. day 1-7 vs 8-14) will be compared between conditions.
  Brachial diastolic blood pressure will be measured with an automated blood pressure monitor (OMRON BP5250).
Weekly average low to high frequency heart rate variability ratio | Immediate post-waking for 14 consecutive days. Weekly averages (e.g. day 1-7 vs 8-14) will be compared between conditions.
  Heart rate variability will be measured with a Polar H10 and the Elite-HRV mobile application.
Weekly averaged Heart rate | Immediate post-waking for 14 consecutive days. Weekly averages (e.g. day 1-7 vs 8-14) will be compared between conditions.
  Heart rate will be measured with a Polar H10 and the Elite-HRV mobile application.

SECONDARY OUTCOMES:
Weekly averaged sleep efficiency | During sleep for 14 consecutive days (7 per condition).
  Wrist-based actigraphy outcome during sleep tracking.
Weekly averaged self-rated sleep quality | Immediate post-waking for 14 consecutive days (7 per condition).
  Self-rated sleep quality on a 5-point Likert scale (1=very poor, 5=very good.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Watso, PhD, Principal Investigator — Florida State University
Locations (1):
- Cardiovascular and Applied Physiology Laboratory, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate data and/or material transfer agreement approvals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after completion of the trial, indefinitely
Access Criteria: A formal plan identifying the intended use of the data and proper completion of appropriate data and/or material transfer agreement approvals with the study PI and their institution.